CLINICAL TRIAL: NCT04552496
Title: The Thyroidectomy Wound Inflammation Can be Caused by Microbes Present in the Thyroid Parenchyma - Observational Research
Brief Title: Cryptic Bacteria of the Thyroid Tissue as a Possible Cause of the Pathology of This Organ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Sergiusz Durowicz, Principal Investigator, Centre of Postgraduate Medical Education
Other Study IDs: 85/PB/2018
Record Dates: First submitted 2020-09-02; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Bacteria Infection Mechanism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presence of cryptic microbes has been widely documented in animal healthy deep tissues.

The thyroid gland is an organ specifically exposed to the microbial environment due to its close location to the mouth microbiome. A number of bacterial phenotypes has been detected in the inflamed thyroid gland. A question raises as to whether bacteria have not already been present in the thyroid gland before the clinical symptoms of goiter became evident.

A problem in thyroid surgery, relatively uncommon but difficult for control, is prolonged thyroidectomy wound healing with skin flap, gland bed inflammation and fibrosis. The causative bacteria may belong to the strains persistently present in the thyroid gland parenchyma. Our objective is to answer questions: a) do the goiter tissue structures contain bacteria, b) if so, which bacterial phenotypes can be identified, c) what are the genetic similarities of the thyroid and periodontal bacterial strains.

Studies are carried out in patients with non-toxic multinodular goiter, toxic multinodular goiter, Graves' disease, single adenoma, Hashimoto's disease, thyroid cancer and recurrent thyroid disease. Tissue harvested during surgery is dissected immediately after thyroidectomy into fragments of parenchyma, arteries, veins and lymph nodes and cultured on Columbia blood agar base for up to 3 weeks. In this method bacteria present in the tissue grow in their natural environment, slowly proliferate and then form the on-plate colonies. It enables detection of even single bacteria usually difficult to be identified in planktonic media. Identification of the isolated bacteria is performed. Their DNA patterns are also compared.

ELIGIBILITY:
Inclusion Criteria:

* thyroid disease requiring surgery

Exclusion Criteria:

* acute or chronic infection at remote sites
* treated with antibiotics over the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with thyroid disease who require surgery. Preoperative clinical diagnosis: 1) non-toxic multinodular goiter, 2) toxic multinodular goiter, 3) Graves disease, 4) single adenoma, 5) Hashimoto's disease, 6) thyroid cancer and 7) recurrent thyroid disease.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
In vivo transferred to ex vivo bacteria culturing in thyroid tissue fragments. The percentage of positive bacterial growth | 30 days
  Thyroid tissue specimens placed on Columbia agar with sheep blood plate and cultured for up to 30 days. Measurement of the percentage of positive bacterial growth.
In vivo transferred to ex vivo bacteria culturing in thyroid tissue fragments. Time lapse to the first bacterial colonies appearance | 30 days
  Thyroid tissue specimens placed on Columbia agar with sheep blood plate and cultured for up to 30 days. Optical assessment of colonies growth kinetic. Measurement of time lapse in days to the first bacterial colonies appearance.
Identification of bacterial strains isolated from cultured thyroid tissue fragments | 3 days
  Isolates identification by standard procedures using the Analytical Profile Identification (API) System (Biomerieux). Assessment of the percentage of bacterial strains cultured from thyroid fragments.
Antibiotic sensitivity of bacterial strains isolated from cultured thyroid tissue fragments | 4 days
  Assessment of the sensitivity of isolated bacterial strains to antibiotics using the ATB system and the ATB-Plus reader (Biomerieux, Paris, France). The percentage of isolated strains sensitive to tested antibiotics.
Isolated bacteria Polymerase Chain Reaction Melting Profiles (PCR MP) | 3 days
  The comparison of DNA patterns of strains isolated from thyroid and oral cavity. The analysis of similarity of the genetic pattern as percentage using the GeneTools program (Syngene, Cambridge, United Kingdom).

CONTACTS AND LOCATIONS:
Overall Officials: Sergiusz Durowicz, MD, PhD, Principal Investigator — Centre of Postgraduate Medical Education, Warsaw, Poland; Marzanna Zaleska, PhD, Principal Investigator — Mossakowski Medical Research Centre, Polish Academy of Sciences, Warsaw, Poland; Waldemar L. Olszewski, MD, PhD, Principal Investigator — Central Clinical Hospital Ministry Interior Administration, Warsaw, Poland; Wiesław Tarnowski, Md, PhD, Principal Investigator — Centre of Postgraduate Medical Education, Warsaw, Poland; Ewa Swoboda-Kopeć, MD, PhD, Principal Investigator — Medical University of Warsaw, Warsaw, Poland
Locations (2):
- Poland (2):
  - Department of General, Oncological and Gastrointestinal Surgery, Centre of Postgraduate Medical Education, Warsaw
  - Department of Applied Physiology, Mossakowski Medical Research Centre, Polish Academy of Sciences, Warsaw